CLINICAL TRIAL: NCT00186875
Title: A Study of Therapy for Pediatric Relapsed or Refractory Acute Lymphoblastic Leukemia
Brief Title: Therapy for Pediatric Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLR17; NCI-2011-01256 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2005-09-01; First posted 2005-09-16 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoma, Lymphoblastic
Keywords: Leukemia; Lymphoblastic; Acute; Lymphoma; Non-Hodgkin's
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Lymphoma | interventions — Etoposide; Cytarabine; Vincristine; Dexamethasone; Methotrexate; Teniposide; pegaspargase; Mitoxantrone; Cyclophosphamide; Mercaptopurine; Vinblastine; Asparaginase; asparaginase erwinia chrysanthemi recombinant; Drug Therapy; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): Participants receive chemotherapy, intrathecal chemotherapy, steroid therapy, hematopoietic stem cell transplant, and natural killer cell transplant as outlined in the Interventions section, including etoposide, cytarabine, vincristine, dexamethasone, methotrexate, teniposide, PEG-asparaginase, mitoxantrone, cyclophosphamide, mercaptopurine, vinblastine, L-asparaginase, erwinia asparaginase.
  Interventions: Drug: Etoposide, cytarabine, vincristine, dexamethasone; Drug: methotrexate, teniposide, PEG-asparaginase; Drug: mitoxantrone, cyclophosphamide, mercaptopurine, vinblastine; Drug: L-asparaginase, erwinia asparaginase; Procedure: chemotherapy, intrathecal chemotherapy, steroid therapy; Procedure: Hematopoietic Stem Cell Transplant; Procedure: Natural Killer (NK) Cell Transplant

INTERVENTIONS:
Drug: Etoposide, cytarabine, vincristine, dexamethasone — See Detailed Description section for details of treatment interventions.
  Other Names: etoposide: VP-16, Vepesid(R); cytarabine: Ara-C, Cytosar-U(R); vincristine: Oncovin(R); dexamethasone: Decadron(R)
Drug: methotrexate, teniposide, PEG-asparaginase — See Detailed Description section for details of treatment interventions.
  Other Names: methotrexate: MTX; teniposide: VM-26, Vumon(R); PEG-asparaginase: Peg-L-Asparaginase, pegaspargase, Oncaspar(R)
Drug: mitoxantrone, cyclophosphamide, mercaptopurine, vinblastine — See Detailed Description section for details of treatment interventions.
  Other Names: mitoxantrone: Novantrone(R); cyclophosphamide: Cytoxan(R); mercaptopurine: 6-MP, Purinethol(R); vinblastine: Velban(R)
Drug: L-asparaginase, erwinia asparaginase — See Detailed Description section for details of treatment interventions.
  Other Names: L-asparaginase: Elspar(R); erwinia asparaginase: Erwinase(R)
Procedure: chemotherapy, intrathecal chemotherapy, steroid therapy — See Detailed Description section for details of treatment interventions.
Procedure: Hematopoietic Stem Cell Transplant — See Detailed Description section for details of treatment interventions.
Procedure: Natural Killer (NK) Cell Transplant — See Detailed Description section for details of treatment interventions.

SUMMARY:
The main purpose of this study is to find out how well participants with relapsed or refractory ALL respond to treatment with an etoposide- and teniposide-based induction chemotherapy regimen and what the side effects are.

Primary Objectives:

* To estimate the response rate for patients with refractory or relapsed ALL.
* To estimate the survival rate of patients with refractory or relapsed ALL treated with risk-directed therapy.

DETAILED DESCRIPTION:
In this study, subjects will be divided into high-risk and standard-risk subgroups according to the length of their first remission, the type of early cancer cell (T or B-cell) and the site or sites of disease relapse. The remission induction phase (the beginning phase of therapy) will consist of three blocks of therapy. Block A features daily IV low-dose etoposide in combination with cytarabine given by continuous IV, weekly vincristine, and daily dexamethasone. In block B, a combination of weekly PEG-asparaginase, vincristine, and daily dexamethasone will be given. Block C will be a combination of high-dose methotrexate, high-dose cytarabine, and teniposide.

There will be two phases of consolidation (treatment phase after induction therapy). Additional therapy will be given between the two consolidation phases. Continuation will consist of eight weekly cycles of chemotherapy. Periodic intrathecal therapy (medicine given into the spinal fluid) will be given throughout the treatment. Participants who do not achieve remission (absence of leukemia) after consolidation will be offered enrollment on St. Jude NKEHM protocol (NK cell transplant). Hematopoietic stem cell transplant (HSCT) is planned for participants with high risk disease. HSCT will be done according to current institutional practice. The duration of chemotherapy will be one year for patients with extramedullary (outside the bone marrow) relapse and two years for all others.

Exploratory objectives include:

* To determine the prevalence of MRD in children undergoing treatment for relapsed ALL and to compare the results to those obtained in children with newly diagnosed ALL.
* To compare the level of MRD in bone marrow and peripheral blood concomitantly in children undergoing treatment for relapsed ALL.
* To characterize the gene expression profile of leukemia cells at the time of diagnosis and relapse to improve our understanding of mechanisms of relapse and of the development of drug resistance.
* To study whether pre-existing or emerging development of serum antibodies to asparaginase is related to hypersensitivity reaction to asparaginase in patient with relapsed ALL.

Detailed Description of Treatment Plan:

All patients will receive the same remission induction. All high-risk patients will be offered HSCT which will be performed after a suitable donor is identified and preferably after MRD becomes negative. If they do not have a donor or they refuse HSCT, they will continue to receive chemotherapy. Standard-risk patients continue chemotherapy if MRD is negative after induction, but will be offered HSCT if MRD is >0.01% after Block C of Induction. Those who do not achieve morphological CR after induction will be treated according to the contingency plan.

Block A (14 days)

Dexamethasone 5 mg/m2/day, days 1-14

Vincristine 1.5 mg/m2 (max 2 mg), days 1 and 8

Etoposide 25 mg/m2, days 1-14

Cytarabine 25 mg/m2, days 1-14

All patients will proceed to Block B if the clinical condition permits.

CNS prophylaxis (IT MHA)

CNS-1: At the time of relapse and day 14.

CNS-2 and 3: At the time of relapse, day 8 and 14.

Leucovorin: 5 mg/m2 (5 mg max dose) PO, 24 and 30 hours after each IT MHA.

Block B (15 days)

All patients will proceed to Block B immediately after Block A if they are clinically well.

Dexamethasone 6 mg/m2, Days 1-14

Vincristine 1.5 mg/m2, days 1 and 8

PEG-Asparaginase 2500 units/m2, days 1, 8 and 15

CNS prophylaxis (IT MHA): CNS-2 or 3 only, if necessary.

* CNS-1: no IT MHA
* CNS-2 and 3: day 8 (minimum 4 doses and maximum 8 doses during induction)

Leucovorin: 5 mg/m2 (5 mg max) PO 24 and 30 hours after each IT MHA

Block C (1 day)

All patients who received Block B will proceed to Block C when WBC >1,000/microL, ANC >300/microL and platelets >50,000 microL after recovery from Block B.

Methotrexate 8 gm/m2, day 1

Cytarabine 1 g/m2 at least 24 h after ITHMA, day 1

Teniposide 165 mg/m2, day 1

CNS prophylaxis (IT MHA):

* CNS-1: at the time of BMA after Block C
* CNS-2 and 3: day 1 and 8 (These two doses of IT MHA may be omitted if the patient had negative CSF for blasts in the 3 preceding CSF exam) and at the time of BMA after Block C (regardless of the previous CSF status).

Leucovorin: 5 mg/m2 (5 mg maximum dose) PO 24 and 30 hours after each IT MHA

Consolidation I

This is a 4-week phase. It will be started if WBC >1000/microL, ANC >500/microL and platelets >50,000 /microL

Week 1: Dex day 1, 2, 3, PEG, VCR, Mito day 4

Week 2: Dex day 1, 2, 3, PEG, VCR, day 4

Week 3: Dex day 1, 2, 3, PEG, VCR, Mito day 4

Week 4: Dex day 1, 2, 3, PEG, VCR, day 4

Dexamethasone 8 mg/m2/day, day 1-3

PEG-Asparaginase 2500 units/m2 IM, day 4 each week

Vincristine 2 mg/m2 (max 2 mg), day 4 each week

Mitoxantrone 12 mg/m2, day 4 week 1 and 3

Interim Continuation

Week 1*†:

etoposide 300 mg/m2 IV, 1 dose on day 1

Cyclophosphamide 300 mg/m2 IV, 1 dose on day 1

Week 2*:

Methotrexate 40 mg/m2 IV, 1 dose on day 1

6-mercaptopurine# 75 mg/m2 PO, Days 1 to 7

Week 3*:

teniposide 150 mg/m2 IV, 1 dose on day 1

Cytarabine 300 mg/m2 IV, 1 dose on day 1

Week 4*:

Dexamethasone§ 12 mg/m2/day PO, TID Days 1 to 5

Vinblastine 6 mg/m2 IV (max 10 mg), 1 dose on day 1

Consolidation II

Week 1*†:

etoposide 300 mg/m2 IV, 1 dose on day 1

Cyclophosphamide 300 mg/m2 IV, 1 dose on day 1

Week 2*:

Methotrexate 40 mg/m2 IV, 1 dose on day 1

6-mercaptopurine# 75 mg/m2 PO, Days 1 to 7

Week 3*:

teniposide 150 mg/m2 IV, 1 dose on day 1

Cytarabine 300 mg/m2 IV, 1 dose on day 1

Week 4*:

Dexamethasone§ 12 mg/m2/day PO, TID, Days 1 to 5

Vinblastine 6 mg/m2 IV (max 10 mg), 1 dose on day 1

Continuation

Week 1*†¶:

etoposide 300 mg/m2 IV, 1 dose on day 1

Cyclophosphamide 300 mg/m2 IV, 1 dose on day 1

Week 2*:

Methotrexate 40 mg/m2 IV, 1 dose on day 1

6-mercaptopurine# 75 mg/m2 PO, QHS, Days 1 to 7

Week 3*:

teniposide 150 mg/m2 IV, 1 dose on day 1

Cytarabine 300 mg/m2 IV, 1 dose on day 1

Week 4:

Dexamethasone§ 12 mg/m2/day PO, TID, Days 1 to 5

Vincristine§ 2 mg/m2 IV(maximum 2mg), 1 dose on day 1

Week 5*‡:

etoposide 300 mg/m2 IV, 1 dose on day 1

Cyclophosphamide 300 mg/m2 IV, 1 dose on day 1

Week 6*:

Methotrexate 40 mg/m2 IV, 1 dose on day 1

6-mercaptopurine# 75 mg/m2 PO, QHS, Days 1 to 7

Week 7*:

teniposide 150 mg/m2 IV, 1 dose on day 1

Cytarabine 300 mg/m2 IV, 1 dose on day 1

Week 8*:

Dexamethasone§ 12 mg/m2/day PO, TID, Days 1 to 5

Vinblastine 6 mg/m2 IV(max 10 mg), 1 dose on day 1

Plan for Stem Cell Transplant

Patients who have positive MRD (high-risk or standard-risk) at the end of induction or all high-risk patients regardless of MRD are eligible for HSCT

* All high-risk patients are eligible for HSCT. HSCT will be performed as soon as MRD becomes negative after induction. If MRD becomes negative (<0.01%) and a donor has not been found, the patient will continue chemotherapy phases (Consolidation I, Interim Continuation, etc) until a suitable donor is found.
* Those who have persistent positive MRD (>0.01%) after Block C are also eligible for HSCT

All standard-risk patients will continue chemotherapy if MRD is negative (<0.01%) after induction.

* If MRD is positive (>0.01%) after Block C of induction, they become eligible for HSCT.
* Standard-risk patients who have no response or progressive disease after Block A and who have positive MRD (>0.01%) after Block B will be candidates for HSCT. They will be re-evaluated after Block C. If MRD after Block C is positive, follow the plan above. If MRD is negative after Block C, the management will be discussed with Transplant Service

Contingency Plan

Patients who do not achieve morphological CR (M1 marrow) after Induction

If CR (M1 marrow) is not achieved after Induction, patients will proceed to Consolidation I. If they do not achieve CR after Consolidation I, they will be offered enrollment on the St. Jude NKHEM protocol or offered alternative therapy. If they do not achieve CR after NKHEM, they will come off treatment.

Patients who achieve CR but have positive MRD (>0.01%) after Block C of induction: Become eligible for HSCT. Up to two more courses of chemotherapy (course 1 and 2) will be given to attempt reducing MRD. They will receive HSCT as soon as MRD becomes negative (MRD may be repeated every 2-4 weeks as indicated).

Standard-risk patients who have positive MRD (>0.01%) after Block B will proceed to Block C. Patients in this category will become candidates for HSCT, but if MRD becomes negative after Block C, the management will be discussed with Transplant Service. Chemotherapy may be administered to reduce MRD prior to HSCT. Patients will be transplanted as soon as the MRD becomes negative.

Patients (high-risk or standard-risk) who achieved CR, but have positive MRD (>0.01%) after Block C of Induction will become eligible for HSCT. Up to two more courses of chemotherapy (course 1 and 2) will be given to attempt reducing MRD. They will receive HSCT as soon as MRD becomes negative. If MRD remains positive after course 2, then, they will proceed to HSCT after discussion with Transplant Service.

Course 1

Give chemotherapy according to the plan for Consolidation I. Start it immediately regardless of CBC. BMA will be performed when WBC >1000/microL, ANC >300/microL and platelets >50,000/microL. If MRD is negative, they will receive HSCT.

Course 2

This course will be given if MRD is positive after Course 1. Patients will be offered enrollment on St. Jude NKHEM protocol.

If they are still MRD positive after Course 2, patients may receive Interim Continuation, Consolidation II, and then Continuation until MRD becomes negative or while awaiting HSCT.

ELIGIBILITY:
Inclusion Criteria

* Childhood ALL in first relapse OR in first hematological relapse after an extramedullary relapse, OR not attaining a complete remission with frontline therapies, OR lymphoblastic leukemia in first relapse.
* Patients must be 21 years of age or younger
* Informed consent explained to and signed by parent/legal guardian.

Exclusion Criteria

* Life expectancy less than 8 weeks
* Patients with mature B cell ALL

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2003-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sima Jeha, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - Rady Children's Hospital and Health Center, San Diego, California
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2004 and August 2012, this study enrolled 47 participants with relapsed or refractory acute lymphoblastic leukemia (ALL): 40 were enrolled at St. Jude and 7 at Rady Children's Hospital.
Pre-assignment Details: Seven participants were excluded from analysis: 6 who enrolled and received treatment prior to a therapy change in amendment 1.0 and one who was incorrectly enrolled on this study. Forty participants were included in the analysis.
Groups:
- Standard Risk: Participants with isolated extramedullary relapse (with blasts in bone marrow (BM) <5%) regardless of the timing of relapse, and participants with B-lineage ALL who develop a late hematological relapse (isolated BM or combined).
- High Risk: Participants with T-cell ALL who develop a hematological [isolated bone marrow (BM) or combined] relapse, irrespective of length of initial remission, participants with B-lineage ALL who develop early hematological relapse (isolated BM or combined), and participants relapsing after hematopoietic stem cell transplantation.
Period: Overall Study
Arm/Group | Standard Risk | High Risk
Started | 26 | 14
Completed | 26 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One patient who was >21 years at diagnosis was enrolled because early versions of the protocol had no upper age limit for participants previously treated on St Jude frontline protocols. The protocol was subsequently amended to change the age criteria to ≤21 years of age at diagnosis for all patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Risk | High Risk | Total
Number analyzed (Participants) | 26 | 14 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.1 (5.0) | 11.3 (6.6) | 11.2 (5.5)
Age, Continuous [Median (Full Range); unit: Years] | 9.7 [3.3 to 22.2] | 12 [2.6 to 21.8] | 10 [2.6 to 22.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 17 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: The "response rate" is defined as the proportion of participants who attain morphological complete remission after the re-induction Block C, inclusive of all patients who begin re-induction. Morphological complete remission was defined as <5% blasts in bone marrow by morphology.
Time Frame: End of re-induction Block C (approximately 1 month after the start of therapy)
Population: Response is defined as morphological complete remission after re-induction Block C. Participants who begin re-induction phase but fail to reach the end of Block C for whatever reason will be regarded as an induction failure.
Measure: Number; unit: proportion of participants
Arm/Group | Standard Risk | High Risk
Number analyzed (Participants) | 26 | 14
proportion of participants
  Complete remission | 0.846 | 0.786
  Failure to reach complete remission | 0.154 | 0.214

2. Primary Outcome: Overall Survival (OS)
Description: OS is measured from the start of on-study to the date of death or to the last date of follow-up. Measurement is determined by Kaplan-Meyer estimate. The probability of survival at 5 years after diagnosis is given.
Time Frame: 2 years after last patient completes therapy (approximately 4 years after enrollment)
Measure: Mean (Standard Deviation); unit: probability
Arm/Group | Standard Risk | High Risk
Number analyzed (Participants) | 26 | 14
probability | 0.654 (0.103) | 0.357 (0.120)

3. Other Pre Specified Outcome: Minimal Residual Disease (MRD) Compared With Historical Data From TOTXV Protocol (NCT00137111)
Description: The prevalence of MRD in children undergoing treatment for relapsed ALL and to compare the results to those obtained in children with newly diagnosed ALL. MRD is considered as positive (i.e., prevalent) if its level is >=0.01%. The prevalence of MRD after Block C is defined as the proportion of MRD positives.
Time Frame: End of Block Block C therapy (Day 46)
Population: Protocol information for the comparison group of TOTXV Participants, including Participant Flow, Baseline Characteristics, and Adverse Events, is available on ClinicalTrials.gov under registration ID NCT00137111.
Measure: Count of Participants; unit: Participants
Groups:
- TOTXV Participants: Total therapy applies to all eligible patients and includes remission induction, consolidation, and continuation therapy. Participants received high-dose methotrexate infusion in upfront window treatment as described in NCT00137111.
Arm/Group | Standard Risk | High Risk | TOTXV Participants
Number analyzed (Participants) | 20 | 9 | 492
Participants
  Negative <0.01% | 11 | 1 | 390
  Positive ≥0.01% | 9 | 8 | 102

4. Other Pre Specified Outcome: Minimal Residual Disease (MRD) Compared With Historical Data From TOTXV Protocol (NCT00137111)
Description: The prevalence of MRD in children undergoing treatment for relapsed ALL and to compare the results to those obtained in children with newly diagnosed ALL. MRD is considered as positive (i.e., prevalent) if its level is >=0.01%. The prevalence of MRD after Block B is defined as the proportion of MRD positives.
Time Frame: End of Block B therapy (Day 19)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Risk | High Risk | TOTXV Participants
Number analyzed (Participants) | 22 | 12 | 488
Participants
  Negative <0.01% | 11 | 2 | 191
  Positive ≥0.01% | 11 | 10 | 297

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time a participant began therapy through 30 days after completion of protocol therapy.
Description: The Other Adverse Events section includes reports of events, Grades 1 through 5.
Arm/Group | Standard Risk | High Risk
Serious Adverse Events (participants affected / at risk) | 6/26 | 2/14
Other Adverse Events (participants affected / at risk) | 26/26 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Risk (N=26) | High Risk (N=14)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0)
Iron overload (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Prolonged QTc interval (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia, supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (3)
Ventricular arrhythmia, ventricular arrhythmia NOS (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 1 (2)
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ulcer, GI, Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI, Stomach (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection, blood (Infections and infestations) | 1 (1) | 1 (1) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L.
Infection, brain (encephalitis, infectious) (Infections and infestations) | 1 (1) | 1 (1) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Infection, Catheter-related (Infections and infestations) | 1 (1) | 0 (0) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Risk (N=26) | High Risk (N=14)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 11 (13) | 0 (0)
Hypertension (Cardiac disorders) | 5 (5) | 3 (3)
Hypotension (Cardiac disorders) | 3 (3) | 3 (5)
Fever (General disorders) | 8 (10) | 0 (0) — In the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L.
Neuroendocrine: ADH secretion abnormality (e.g., SIADH or low ADH) (Endocrine disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (3) | 2 (2)
Mucositis/stomatitis (clinical exam), oral cavity (Gastrointestinal disorders) | 3 (9) | 0 (0)
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Febrile neutropenia (General disorders) | 17 (29) | 7 (11) — Fever of unknown origin without clinically or microbiologically documented infection (ANC <1.0 x 10e9/L).
Infection, blood (Infections and infestations) | 9 (11) | 2 (2) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Infection, sinus (Infections and infestations) | 7 (8) | 0 (0) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 6 (9) | 0 (0)
Infection, catheter-related (Infections and infestations) | 3 (3) | 3 (3) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Infection with normal ANC or Grade 1 or 2 neutrophils, upper airway NOS (Infections and infestations) | 6 (8) | 0 (0)
Infection, lung (pneumonia) (Infections and infestations) | 4 (4) | 1 (1)
Infection, upper airway NOS (Infections and infestations) | 4 (4) | 0 (0) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Infection, skin (cellulitis) (Infections and infestations) | 3 (3) | 1 (1) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Infection with normal ANC or Grade 1 or 2 neutrophils, skin (cellulitis) (Infections and infestations) | 4 (6) | 1 (1)
Infection, other (Infections and infestations) | 1 (1) | 3 (4)
Infection, pharynx (Infections and infestations) | 2 (2) | 0 (0) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Infection with normal ANC or Grade 1 or 2 neutrophils, lung (pneumonia) (Infections and infestations) | 2 (2) | 0 (0)
Infection, lip/perioral (Infections and infestations) | 1 (1) | 1 (1) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Infection, wound (Infections and infestations) | 1 (1) | 1 (1) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L).
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 8 (10) | 6 (11)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 9 (12) | 4 (6)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (6) | 5 (7)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 (7) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
Amylase (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Lipase (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Neuropathy, motor (Nervous system disorders) | 5 (5) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Neuropathy, sensory (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (2) | 1 (1)
Pain, neuralgia/peripheral nerve (General disorders) | 8 (8) | 1 (1)
Pain, extremity-limb (General disorders) | 5 (5) | 1 (1)
Pain, back (General disorders) | 4 (7) | 0 (0)
Pain, abdomen NOS (General disorders) | 2 (2) | 0 (0)
Pain, head/headache (General disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (4) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes